CLINICAL TRIAL: NCT00117936
Title: Human Recombinant Fibroblast Growth Factor-1 (FGF-1), for the Treatment of Subjects With Severe Coronary Heart Disease, a Placebo Controlled, Double-blind, Dose-varying Study
Brief Title: Fibroblast Growth Factor-1 (FGF-1) for the Treatment of Coronary Heart Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CardioVascular BioTherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CVBT-CHD07-01; NCT00032318 (obsolete NCT alias)
Record Dates: First submitted 2005-06-30; First posted 2005-07-11 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Coronary Disease; Coronary Heart Disease; Myocardial Ischemia; Coronary Arteriosclerosis
Keywords: Angiogenesis; No-option heart patients; Blocked coronary artery; Revascularization; FGF-1; growth factor
MeSH Terms: conditions — Coronary Disease; Myocardial Ischemia; Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (3):
- 1 (Experimental): Human Recombinant Fibroblast Growth Factor-1 (FGF 1-141) - high dose, given as intramyocardial injections via a NOGA Injection Catheter, single cath lab session.
  Interventions: Combination Product: Human Recombinant Fibroblast Growth Factor-1 (FGF 1-141) - low dose
- 2 (Experimental): Human Recombinant Fibroblast Growth Factor-1 (FGF 1-141) - low dose, given as intramyocardial injections via a NOGA Injection Catheter, single cath lab session.
  Interventions: Combination Product: Human Recombinant Fibroblast Growth Factor-1 (FGF1-141) - high dose
- 3 (Placebo Comparator): Placebo solution void (not containing) Human Recombinant Fibroblast Growth Factor-1 (FGF 1-141), given as intramyocardial injections via a NOGA Injection Catheter, single cath lab session.
  Interventions: Combination Product: Placebo

INTERVENTIONS:
Combination Product: Human Recombinant Fibroblast Growth Factor-1 (FGF 1-141) - low dose — Up to ten intramyocardial injections of low dose FGF 1-141, via a NOGA Injection Catheter, single cath lab session
  Arms: 1
Combination Product: Human Recombinant Fibroblast Growth Factor-1 (FGF1-141) - high dose — Up to ten intramyocardial injections of high dose group (FGF-1-141), via a NOGA Injection Catheter, single cath lab session
  Arms: 2
Combination Product: Placebo — Up to ten intramyocardial injections of placebo via a NOGA Injection Catheter, single cath lab session
  Arms: 3

SUMMARY:
Treatment for no-option heart patients with coronary artery disease. Procedure includes the injection into the heart of a protein growth factor, administered by the Biological Delivery Systems MyoStar injection and mapping catheters, to stimulate the growth of blood vessels around blocked coronary arteries.

DETAILED DESCRIPTION:
Patients with chronic, stable angina with documented coronary artery disease are eligible for the study.

ELIGIBILITY:
Inclusion criteria

1. Sign an informed consent form.
2. Age ≥25 and ≤75 years, either gender, and any race.
3. At least a 3 month history of chronic, stable angina and is relieved by rest and/or nitroglycerin.
4. Documented symptomatic CCS Angina Classification of III to IV despite use of optimal medical therapy as noted in Inclusion Criterion 10.
5. Pattern of CHD (coronary pathology) where percutaneous interventional therapy and/or CABG is not recommended by the treating cardiologist. This decision should have a documented basis in either complicated vessel physiology and/or lack of suitable target vessels for both PTCA and CABG, or past history of complications.
6. One/two/three vessel disease as evidenced either by an angiographic documentation of advanced atherosclerotic narrowing of ≥60% of at least one major epicardial coronary artery (right coronary artery [RCA], left circumflex [LCX], or LAD [or any of their branches]), or of diffuse type of CHD as evidenced by the appearance on coronary angiography of multiple stenoses, multiple atherosclerotic plaques, and/or peripheral occlusion(s) of coronary vessel(s) with and without a history of MIs.
7. demonstrate a radionuclide or angiographically determined left ventricular ejection fraction (LVEF) ≥30%.
8. Pre-operative proof of reversible ischemia.
9. No evidence of proliferative retinopathy or significant non-proliferative retinopathy.
10. must be on optimal medical therapy for at least 2 months prior to entering the study, as documented by a medical history. This will include medical management, and subjects must enter the study on at least one of the following medications: beta-blockers, calcium entry blockers, ranolizine, or long-acting nitrates.
11. Exercise duration during the qualifying treadmill tests at Visit 1 and Visit 2 is ≥3 and ≤9 minutes on a modified Bruce protocol.
12. Exercise durations for the qualifying treadmill tests at Visits 1 and 2 must satisfy at least one of the two following conditions: (a) they differ by less than or equal to 20% of the longer time; (b) they differ by less than or equal to 60 seconds. Subjects whose ETTs at Visits 1 and 2 do not satisfy at least one of these two conditions are allowed a third ETT, at the investigator's discretion, from 5 to 7 days after Visit 2. If a third ETT is done, then when compared with the second ETT it must satisfy at least one of the two conditions above.
13. For a treadmill test result to support inclusion it must terminate in the presence of angina for either of the following reasons: (a) angina becomes too severe to continue the test AND there must be a horizontal depression or downsloping ST-segment of at least 1 mm measured 80 ms from the J point as subsequently established by the Biomedical Systems central ECG lab, or (b) angina of any grade AND there must be a horizontal depression or downsloping ST-segment measured 80 ms from the J point of 2 mm during exercise. The qualifying time for the treadmill test will then be the time to a horizontal depression or downsloping ST-segment of 1 mm compared to the pre-exercise ST segment as subsequently established by the Biomedical Systems central ECG lab.
14. A forced vital capacity (FVC) of ≥30%.
15. A negative pregnancy test in women of childbearing potential at Screening.
16. Female subjects must be post-menopausal or sterilized, or if she is of childbearing potential, she is not breast feeding, has no intention to become pregnant during the course of the study, and is using contraceptive drugs or devices.
17. Negative cancer screening tests according to the American Cancer Society ([ACS] Appendix 13.8).
18. Ability to complete the study in compliance with the protocol.

Exclusion criteria

1. History of undergoing a CABG, PTCA or TMR or evidence of an acute MI in the last 3 months.
2. Subjects with malignancies or a history of malignancies (with the exception of basal cell carcinoma [BCC] of the skin) will be excluded from the study. Those subjects with a history of BCC are eligible for enrollment, and will be monitored by a qualified dermatologist every 8 weeks for a period of 6 months for evaluation of their skin condition. Subjects with existing BCC will be excluded from the study.
3. Evidence of concurrent clinically significant infection (e.g. elevated white blood cell [WBC] count >13,000 x 109/L, temperature >38.5°C), evidence of "common cold" or "flu."
4. Concomitant other structural heart disease, such as moderate to severe heart valve disease, congenital heart disease, etc. other than evidence of congestive heart failure that is directly related to past ischemic events.
5. Left ventricular thrombus (mobile or mural-based) as evidenced by ventriculogram or echocardiography.
6. Creatine kinase (CK) levels >3 x upper limit of normal (ULN).
7. Renal insufficiency requiring dialysis or laboratory evidence of a serum creatinine >2.0 mg/dL.
8. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2 x ULN.
9. History of coagulation disorders or abnormal prothrombin time (PT) or partial thromboplastin time (PTT) >1.5 x ULN, thrombocytopenia (<100,000/µl), or ongoing anticoagulant therapy (with the exception of aspirin, up to 85 mg/day).
10. History of blood cell diseases.
11. Poorly controlled insulin-dependent diabetes mellitus (HbA1c >8%)
12. Pre-existing retinal disease, including proliferative retinopathy, severe nonproliferative retinopathy.
13. Use of any illicit recreational drugs within the past year.
14. A positive test result for human immunodeficiency virus (HIV) antibody.
15. Screening ECG results demonstrating recent evidence of transmural ischemia.
16. Clinically significant ECG abnormalities, e.g.: QRS duration >0.12 seconds; QTc >450 ms in males or >460 ms in females;High-grade trioventricular (AV) block; Left bundle branch block(LBBB; Left ventricular hypertrophy(LVH) with secondary ST-T changes; Frequent, recurrent, or sustained ventricular arrhythmia; Resting ST segment depression >1 mm (measured 80 ms beyond the J point) at baseline.
17. Subjects having a concomitant life-threatening disease in which their life expectancy is estimated to be less than 2 years.
18. Any condition which in the opinion of the investigator would interfere with the participant's ability to provide informed consent and comply with study instructions, possibly confound interpretation of study results, or endanger the participant if he took part in the trial.
19. Use of an investigational drug, device or product, or participation in a drug research study within a period of 30 days prior to receiving IMP.
20. Any subject with unstable angina.
21. Heart failure New York Heart Association (NYHA) Functional Class III or IV.
22. Uncontrolled hypertension precluding exercise testing and/or contributing to angina severity (systolic blood pressure [SBP] >200 mmHg or diastolic blood pressure [DBP] >110 mmHg), or significant hypotension (SBP <90 mmHg or DBP <60 mmHg).
23. Subjects currently on External Counter Pulsation therapy or who have received this therapy within 3 months prior to the screening date.
24. Any mobility or pulmonary complication that impedes the subject's ability to perform an exercise stress test.
25. Total fasting serum cholesterol >200 mg/dL (if levels greater than or equal to 200 mg/dL, additional medical interventions can be initiated to bring levels below 200 mg/dL).
26. History of heparin-induced thrombocytopenia.
27. Subjects with a history of recurrent symptomatic atrial fibrillation or significant ventricular arrhythmias.
28. Aortic or mitral valve replacement.
29. Subjects who have undergone heart transplantation.
30. Medical history and physical examination displaying any evidence that catheterization is contraindicated.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Change in cardiac perfusion as measured by cMRI scan under stress conditions and change in vascular bed density at the sites of injections as determined by angiography | 1 year
  Change in cardiac perfusion as measured by cMRI scan under stress conditions and change in vascular bed density at the sites of injections as determined by angiography
Change in CCS angina score | baseline to 12 weeks, followed up to one year
  Change in CCS angina score

SECONDARY OUTCOMES:
Exercise treadmill test: time (or change in time) to onset of at least 1 mm additional horizontal or downsloping ST-segment depression, or time to ETT in the absence of at least 1 mm additional ST-segment depression due to pain (angina) | 1 year
  Exercise treadmill test: time (or change in time) to onset of at least 1 mm additional horizontal or downsloping ST-segment depression, or time to ETT in the absence of at least 1 mm additional ST-segment depression due to pain (angina)

CONTACTS AND LOCATIONS:
Overall Officials: Emerson Perin, MD, PhD, Principal Investigator — Texas Heart Institute

REFERENCES:
- See also: web site of sponsor — http://www.cvbt.com